CLINICAL TRIAL: NCT00032032
Title: Phase I/II Study Of Concurrent Chemotherapy And Escalating Doses Of Radiotherapy (RT) For Unresectable Non-Small Cell Lung Cancer (NSCLC) Using A New RT Paradigm
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0028; NCI-2012-02458 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000069250 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy + paclitaxel + carboplatin (Experimental): Patients undergo radiotherapy once daily 5 days a week for 7 weeks and 2 days (a total of 37 fractions). Patients concurrently receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes once weekly for 7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Beginning 3 weeks after completion of radiotherapy, patients receive paclitaxel and carboplatin as above. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, once during the last week of radiotherapy, and then every 3 months for 2 years.
  Patients are followed at 3 weeks, every 3 months for 21 months, and then every 6 months for 3 years.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of radiation therapy when given with combination chemotherapy and to see how well they work in treating patients with non-small cell lung cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of radiotherapy in combination with carboplatin and paclitaxel in patients with unresectable non-small cell lung cancer.
* Determine the 2-year survival of patients treated with this regimen.
* Determine the progression-free local control rate in patients treated this regimen.
* Determine the tolerability of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of radiotherapy.

Patients undergo radiotherapy* once daily 5 days a week for 7 weeks and 2 days (a total of 37 fractions). Patients concurrently receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes once weekly for 7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

NOTE: *No prophylactic nodal radiotherapy is administered

Cohorts of 3-6 patients receive escalating doses of radiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 12 additional patients are treated at that dose level in the phase II portion of the study.

Beginning 3 weeks after completion of radiotherapy, patients receive paclitaxel and carboplatin as above. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, once during the last week of radiotherapy, and then every 3 months for 2 years.

Patients are followed at 3 weeks, every 3 months for 21 months, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage I, II, or III NSCLC that is unresectable due to tumor extent or other medical reasons
* Measurable disease
* Tumor must not exceed volume that would require radiation volumes greater than those allowed on this study
* No more than blunting of the costophrenic angle on chest x-ray due to pleural effusions
* No more than small effusions seen on chest CT scan only
* No supraclavicular adenopathy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Total bilirubin no greater than 1.5 times upper limit of normal (ULN) OR
* Direct bilirubin no greater than 1.5 times ULN
* AST no greater than 3 times ULN

Renal:

* Creatinine clearance at least 40 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* FEV_1 at least 1 L or 35% of predicted

Other:

* No grade 2 or greater peripheral neuropathy
* No weight loss of 10% or more within the past 3 months
* No uncontrolled infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinoma (carcinoma in situ), or localized prostate cancer
* No other severe underlying disease that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic:

* No prior biologic therapy for NSCLC
* No concurrent biologic therapy
* No concurrent prophylactic filgrastim (G-CSF)

Chemotherapy:

* No prior chemotherapy for NSCLC
* No other concurrent chemotherapy

Endocrine therapy:

* No prior endocrine therapy for NSCLC

Radiotherapy:

* No prior radiotherapy for NSCLC

Surgery:

* No prior surgery for NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2002-05; Primary Completion 2008-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) as assessed by dose-limiting toxicity within 1 month after completion of study treatment (phase I) | Up to 1 month
Survival at 2 years (phase II) | Up to 2 years

SECONDARY OUTCOMES:
Survival time | Up to 5 years
Toxicity | Up to 5 years
Time to progression | Up to 5 years
Time to local progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Schild, MD, Study Chair — Mayo Clinic
Locations (51):
- United States (51):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - McFarland Clinic, PC, Ames, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin

REFERENCES:
- [Result] Schild S, Graham D, Hillman S, et al.: Survival of patients (pts) treated with high-dose radiotherapy (RT) and concurrent chemotherapy for unresectable non-small cell lung cancer (NSCLC). [Abstract] J Clin Oncol 27 (Suppl 15): A-7544, 2009.
- [Result] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Derived] Schild SE, Hillman SL, Tan AD, Ross HJ, McGinnis WL, Garces YA, Graham DL, Adjei AA, Jett JR; Mayo Clinic, North Central Cancer Treatment Group. Long-Term Results of a Trial of Concurrent Chemotherapy and Escalating Doses of Radiation for Unresectable Non-Small Cell Lung Cancer: NCCTG N0028 (Alliance). J Thorac Oncol. 2017 Apr;12(4):697-703. doi: 10.1016/j.jtho.2016.12.021. Epub 2017 Jan 12. PMID 28089762